CLINICAL TRIAL: NCT05583318
Title: Living Conditions After Non-Hodgkin's Lymphoma in France
Acronym: LymphoVie 2
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: MAYNADIE 2022
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Non-hodgkin's Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Data Collection; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Part 1: Patients diagnosed with non-Hodgkin's lymphoma: Diagnosis period 2010-2018, from the hematological malignancy registries of Côte-d'Or, Gironde, Basse-Normandie
  Interventions: Other: Data collection
- Part 2: Patients diagnosed with live non-Hodgkin's lymphoma after vital status update: Update of vital status in December 2022
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Data collection — Data from hematological malignancy registries
  Groups: Part 1: Patients diagnosed with non-Hodgkin's lymphoma
Other: Questionnaires — 9 questionnaires were sent out:
  1. QLQ-C30 and SF-12 Quality of Life Questionnaire.
  2. Oral quality of life questionnaire QLQ-OH15
  3. Sexuality questionnaire SHQ-C22
  4. Anxiety and depression questionnaire HADS,
  5. Rosenberg Self-Esteem Questionnaire
  6. RNLI Reintegration to Normal Life Questionnaire
  7. Social Support Questionnaire SSQ6,
  8. Socio-economic status questionnaire EPICES,
  9. Complementary questionnaire collecting data on socio-professional status.
  Groups: Part 2: Patients diagnosed with live non-Hodgkin's lymphoma after vital status update

SUMMARY:
This is an innovative project, allowing to study for the first time the long-term living conditions of patients after diffuse large B-cell lymphoma (DLBCL) or follicular lymphoma (FL) from population data in France. Patients will be selected from the three specialized hematology registries in France: Côte-d'Or, Gironde and Basse-Normandie.

This is also one of the first studies to look at epidemiological indicators of net survival after diagnosis of follicular lymphoma and diffuse large B-cell lymphoma, adjusted for clinical factors such as disease stage, therapeutic management, and comorbidities, apart from the standard adjustment factors of age, sex, and time of diagnosis in real life. In addition, the proportion of cured patients will be estimated.

For component 1, this will be the survival analysis on the initial data. For part 2, questionnaires will be sent out followed by a follow-up if necessary one month after the mailing. There is no physical interview nor any specific biological or imaging examination.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis period 2010-2018, according to the 2008 WHO ICD-O-3 classification, from the hematological malignancy registries of Côte-d'Or, Gironde, Basse-Normandie
* Patients with a diagnosis of follicular lymphoma (9690/3, 9691/3, 9695/3, 9698/3, 9597/3)
* Patients with a diagnosis of diffuse large B-cell lymphoma (9678/3, 9679/3, 9680/3, 9684/3, 9688/3, 9712/3, 9735/3, 9737/3, 9738/3)
* For Part 2: Individuals alive at the date of vital status update

Non-inclusion criteria:

* Other forms of malignant hemopathies at diagnosis,
* Minors.

Exclusion Criteria:

* Person under a legal protection measure (curatorship, guardianship)
* Person under a legal protection measure (guardianship, tutorship)
* Pregnant, parturient or breastfeeding women
* Major incapable or unable to express his consent
* Person who did not return the questionnaires following the 1-month follow-up, or patient who expressed refusal to participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-Hodgkin's lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 1570 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | December 2022
  Update of vital status (part 1)
Generic SF-12 questionnaire | October 2024
  Mesure of the quality of life (part 2)
Specific QLQ-C30 questionnaire | October 2024
  Mesure of the quality of life (part 2)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: No